CLINICAL TRIAL: NCT02433080
Title: Randomised, Controlled, Pilot Clinical Trial to Assess the Feasibility of a Healthy Eating and Physical Activity Program in Endometrial Cancer Survivors
Brief Title: Diet and Physical Activity in Uterine Cancer Survivors
Acronym: DEUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14/0765
Record Dates: First submitted 2015-04-20; First posted 2015-05-04 (Estimated); Results first posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Endometrial Neoplasms
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shape-Up following cancer treatment (Active Comparator): In addition to usual care, cancer survivors in the intervention group will participate in a behaviour change programme, called "Shape-Up following cancer treatment: a self-help programme on eating well and being active". Participants will be allocated to groups of eight to ten. These groups will meet every week for eight weeks and each session will last approximately 90 minutes. The programme focuses on strategies for improving diet and physical activity in a self-help and peer education format. Each week, one participant will volunteer to present a new concept (e.g. regular eating, being active, eating a balanced diet, keep an eye on portion sizes, and manage internal and external triggers, and understanding food labeling) to the rest of the group.
  Interventions: Behavioral: Shape-Up following cancer treatment
- Control intervention (No Intervention): Participants in the control group will be offered usual care until the 24-week follow-up. Quantifying usual care is challenging, but preliminary qualitative work suggested that most survivors do not received any unsolicited advice about healthy eating and physical activity from their health care professionals after treatment.
  During the course of their participation in the trial, participants will be contacted only for the assessments. After the completion of the 24-week follow-up, participants will receive the booklet "Healthy living after cancer"; a brief self-help manual produced by the World Cancer Research Fund. Providing only this information aims to match the currently offered usual care as accurately as possible but also meet ethical standards.

INTERVENTIONS:
Behavioral: Shape-Up following cancer treatment — The programme is based on "Social Cognitive Theory" and "Control Theory". The focus of the programme lies on self-control, self-efficacy, and relapse prevention.
  Other Names: Self-help healthy eating and physical activity programme
  Arms: Shape-Up following cancer treatment

SUMMARY:
Endometrial cancer is the most common gynaecological cancer in developed countries with more than 75% of the patients surviving for at least five years. However, most endometrial cancer survivors are overweight and obese and do not meet the current nutrition and physical activity recommendations. This can lower their quality of life and increase their risk for chronic diseases. Behaviour change interventions can help them feel better about themselves and improve their quality of life. Applying them shortly after treatment seems ideal as cancer survivors feel motivated to make changes about their lifestyle at this time point.

This study is to see if the investigators can design a project to measure how well a psycho-educational healthy eating and physical activity programme tailored to the survivors' needs works. Sixty-four endometrial cancer survivors diagnosed during the previous three years, and are all clear will be put by chance into one of two groups. One will receive the program. The other will receive usual care until the end of the trial and, then, a discussion and a self-help guide about eating well and being active following cancer treatment. This will help us to see if the programme makes a difference compared with usual care. The results will inform a larger study to test if a lifestyle program can improve the quality of life of uterine cancer survivors compared with usual care. The investigators will change the programme materials in response to the investigators' findings, making them available to services. The results will inform practice and research.

DETAILED DESCRIPTION:
Low physical activity, poor diet and obesity are risk factors for the development of endometrial cancer. A growing body of evidence suggests that they may be linked with quality of life after cancer treatment. However, only about 1% of endometrial cancer survivors seem to meet the current fruit and vegetable, physical activity, and non-smoking recommendations; while 57% meets only the non-smoking recommendations, and 22% meet none of the recommendations,

These behaviours exist despite cancer diagnosis being perceived as a "teachable moment". Capitalising the "teachable moment" of cancer, behaviour change interventions in high-risk populations might be more effective than those targeting the general population.

Theory-based behaviour change interventions suggest that improving diet and physical activity is safe, acceptable, and feasible and can help cancer survivors improve their quality of life. In contrast, there are only limited studies to support these data in the United Kingdom to allow generalisability of these results. However, the majority of these interventions were long-term and resource intensive which may render them inappropriate for wide dissemination. Therefore, feasible and effective interventions are needed to promote implementation of the nutrition and physical activity guidelines.

The intervention is based on the Shape-Up eight-week weight management programme. This programme is based on "Social Cognitive Theory" and "Control Theory". A version of this program has been favourably evaluated in terms of acceptability, physical, and psychological outcomes. We have tailored this programme (Shape-Up following cancer treatment) to help endometrial cancer survivors improve their diet, and activity pattern. The focus of the programme lies on self-control, self-efficacy, and relapse prevention in terms of healthy eating and physical activity. Behavioural techniques will include self-monitoring of behaviour with the use of food and physical activity diaries, behavioural goal setting, action planning, graded tasks, problem solving, self-reward, and review of behavioural goals. It will also provide information about health consequences and emotional consequences, pros and cons, behavioural practice, habit formation, reducing exposure to cues for the behaviour, behaviour substitution, distraction, social support (unspecified), demonstration of behaviour (for resistance exercises), instructions on how to perform the behaviour (for resistance exercises), and reframing.

The DEUS pilot trial is an eight-week, two-arm, individually randomised, controlled pilot trial comparing the use of the "Shape-Up following cancer treatment" programme to usual care. According to Medical Research Council guidance for complex interventions, this is a Phase 2 feasibility study. Randomisation will be performed with minimisation using a 1:1 allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged >18 years (no upper age limit)
2. Women diagnosed with endometrial cancer (C54.1) within the previous 36 months
3. Women who are able to understand spoken and written English

Exclusion Criteria:

1. Women with stage IVB (metastatic) endometrial cancer (any metastasis beyond the pelvis)
2. Women on active anti-cancer, and/or palliative treatment,
3. Women having second primary cancer
4. Women who lack mental capacity to decide to take part in the study and to participate in it (upon clinical team's judgement in accordance with the Mental Capacity Act 2005 Code of Practice 2007)
5. Women with severe depression (upon consultant's judgement based on the Diagnostic and Statistical Manual of Mental Disorders-IV criteria)
6. Women unavailable for longitudinal follow-up assessments
7. Women who participated in a professionally delivered weight loss or exercise program during the previous 6 months
8. Women with a World Health Organization performance score 3-4

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Lanceley, PhD, Principal Investigator — University College, London
Locations (2):
- United Kingdom (2):
  - Barts Health NHS Trust, London, Greater London
  - University College London Hospital NHS Trust, London, Greater London

REFERENCES:
- [Background] Chiuve SE, Fung TT, Rimm EB, Hu FB, McCullough ML, Wang M, Stampfer MJ, Willett WC. Alternative dietary indices both strongly predict risk of chronic disease. J Nutr. 2012 Jun;142(6):1009-18. doi: 10.3945/jn.111.157222. Epub 2012 Apr 18. PMID 22513989
- [Background] Koutoukidis DA, Lopes S, Atkins L, Croker H, Knobf MT, Lanceley A, Beeken RJ. Use of intervention mapping to adapt a health behavior change intervention for endometrial cancer survivors: the shape-up following cancer treatment program. BMC Public Health. 2018 Mar 27;18(1):415. doi: 10.1186/s12889-018-5329-5. PMID 29587699
- [Derived] Koutoukidis DA, Beeken RJ, Manchanda R, Burnell M, Ziauddeen N, Michalopoulou M, Knobf MT, Lanceley A. Diet, physical activity, and health-related outcomes of endometrial cancer survivors in a behavioral lifestyle program: the Diet and Exercise in Uterine Cancer Survivors (DEUS) parallel randomized controlled pilot trial. Int J Gynecol Cancer. 2019 Mar;29(3):531-540. doi: 10.1136/ijgc-2018-000039. Epub 2019 Feb 4. PMID 30723098
- [Derived] Koutoukidis DA, Beeken RJ, Manchanda R, Michalopoulou M, Burnell M, Knobf MT, Lanceley A. Recruitment, adherence, and retention of endometrial cancer survivors in a behavioural lifestyle programme: the Diet and Exercise in Uterine Cancer Survivors (DEUS) parallel randomised pilot trial. BMJ Open. 2017 Oct 8;7(10):e018015. doi: 10.1136/bmjopen-2017-018015. PMID 28993394
- [Derived] Koutoukidis DA, Beeken RJ, Manchanda R, Burnell M, Knobf MT, Lanceley A. Diet and exercise in uterine cancer survivors (DEUS pilot) - piloting a healthy eating and physical activity program: study protocol for a randomized controlled trial. Trials. 2016 Mar 10;17(1):130. doi: 10.1186/s13063-016-1260-1. PMID 26965165

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 60 participants were enrolled, only 54 were included in the study analysis as the remaining 6 participants were deemed ineligible to participate and excluded from the analysis.
Period: Overall Study
Arm/Group | Shape-Up Following Cancer Treatment | Control Intervention
Started | 26 | 28
8 Weeks | 25 | 24
Completed (24 weeks and analyzed) | 25 | 24
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Shape-Up Following Cancer Treatment | Control Intervention | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (9) | 61.5 (7.7) | 62.1 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 25 | 24 | 49

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rate (Percentage of Potentially Eligible Participants Who Were Enrolled to the Study)
Description: Achieving a 30% recruitment rate of the potentially eligible participants
Time Frame: 6 months
Population: Of the 296 potentially eligible participants, 20.3% were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Both Arms Combined: Recruitment to the trial overall
Arm/Group | Both Arms Combined
Number analyzed (Participants) | 296
percentage of participants | 20.3 [15.7 to 24.9]

2. Secondary Outcome: Change From Baseline in Health-related Quality of Life Score
Description: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 & European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Endometrial Cancer Module 24 Global quality of life scale ranging from 0-100 with higher scores indicating better quality of life
Time Frame: Baseline, 8weeks, 24weeks
Measure: Mean (Standard Deviation); unit: units on the global QoL scale 0-100
Arm/Group | Shape-Up Following Cancer Treatment | Control Intervention
Number analyzed (Participants) | 25 | 24
units on the global QoL scale 0-100
  8week change from baseline | 3.0 (11.3) | 8.7 (14.5)
  24week change from baseline | 8.7 (14.5) | -1.4 (14.7)
Statistical Analysis 1: Comparison: Shape-Up Following Cancer Treatment vs Control Intervention; This statistical analysis applies for the outcomes 2-8; Test type: Other; p = 0.05, ANCOVA; Mean Difference (Net) = 6.4, 95% CI 2-sided [-3.6 to 16.5]

3. Secondary Outcome: Change From Baseline in Dietary Quality (24-h Dietary Recall)
Description: One 24-h dietary recall for each timepoint. This is the combined total Alternate healthy eating index-2010 score ranging from 0-110 with higher scores indicating higher dietary quality.
Time Frame: Baseline, 8weeks, 24weeks
Population: The outcome measure values below refer to the change at 24weeks from baseline using an ANCOVA model
Measure: Mean (Standard Deviation); unit: units on a scale (AHEI-2010)
Arm/Group | Shape-Up Following Cancer Treatment | Control Intervention
Number analyzed (Participants) | 25 | 24
units on a scale (AHEI-2010)
  8week change from baseline | 4.4 (15.3) | -2.9 (14.1)
  24week change from baseline | 3.0 (14.0) | 2.2 (17.8)

4. Secondary Outcome: Change From Baseline in Physical Activity (Physical Activity Recall)
Description: 7-day physical activity recall
Time Frame: Baseline, 8weeks, 24weeks
Measure: Mean (Standard Deviation); unit: MET-h/day
Arm/Group | Shape-Up Following Cancer Treatment | Control Intervention
Number analyzed (Participants) | 25 | 24
MET-h/day
  8week change from baseline | -1.4 (2.2) | -1.8 (3.6)
  24week change from baseline | 0.2 (2.1) | 0.4 (2.7)

5. Secondary Outcome: Change From Baseline in Hand-grip Strength
Time Frame: Baseline, 8weeks, 24weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Shape-Up Following Cancer Treatment | Control Intervention
Number analyzed (Participants) | 25 | 24
kg
  8week change from baseline | -0.3 (2.4) | -1.7 (3.1)
  24week change from baseline | 0.0 (2.4) | -1.3 (1.9)

6. Secondary Outcome: Change From Baseline in Weight
Time Frame: Baseline, 8weeks, 24weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Shape-Up Following Cancer Treatment | Control Intervention
Number analyzed (Participants) | 25 | 24
kg
  8week change from baseline | -0.9 (1.1) | 0.3 (1.5)
  24week change from baseline | -1.1 (2.6) | -0.2 (2.5)

7. Secondary Outcome: Change From Baseline in Fat Mass Index
Description: Using MC980 multi-frequency segmental body composition analyser. Fat mass index was calculated as kg of fat mass divided by squared height in meters.
Time Frame: Baseline, 8weeks, 24weeks
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Shape-Up Following Cancer Treatment | Control Intervention
Number analyzed (Participants) | 25 | 24
kg/m2
  8week change from baseline | -0.1 (0.8) | 0.1 (0.5)
  24week change from baseline | -0.4 (0.8) | -0.2 (0.8)

8. Secondary Outcome: Intervention Evaluation Questionnaire
Description: Change in the self-assessment of the gained skills (Shape-Up self-efficacy score). This is a total score 0-5 with higher scores indicating higher self-efficacy.
Time Frame: 8weeks, 24weeks
Population: Missing data for 2 people in the Shape-up group
Measure: Mean (Standard Deviation); unit: units on a scale 0-5
Arm/Group | Shape-Up Following Cancer Treatment | Control Intervention
Number analyzed (Participants) | 25 | 24
units on a scale 0-5
  8week change from baseline: number analyzed (Participants) | 23 | 24
  8week change from baseline | 0.2 (0.5) | -0.2 (0.7)
  24week change from baseline: number analyzed (Participants) | 23 | 24
  24week change from baseline | 0.1 (0.5) | -0.1 (0.3)

9. Secondary Outcome: Health Care Services Use - Medication
Description: Number of currently prescribed medications over the 24 weeks of the trial (Self-reported)
Time Frame: 24weeks
Measure: Mean (Standard Deviation); unit: Prescribed medications
Arm/Group | Shape-Up Following Cancer Treatment | Control Intervention
Number analyzed (Participants) | 25 | 24
Prescribed medications | 1.4 (2.2) | 1.5 (1.7)

10. Secondary Outcome: Adherence Rate
Description: The percentage of engaged participants attending at least one of the last three sessions of the intervention. Engaged participants are those who have attended at least two sessions of the intervention.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Shape-Up Following Cancer Treatment
Number analyzed (Participants) | 26
Participants | 20

11. Secondary Outcome: Retention Rate
Description: Rate of complete follow-up
Time Frame: Baseline to 24weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Shape-Up Following Cancer Treatment | Control Intervention
Number analyzed (Participants) | 26 | 28
Participants | 25 | 24

12. Secondary Outcome: Health Care Services Use - Number of General Practitioner Visits
Description: Number of visits to their general practitioner over the 24 weeks of the trial (Self-reported)
Time Frame: 24weeks
Measure: Mean (Standard Deviation); unit: Visits to the general practitioner
Arm/Group | Shape-Up Following Cancer Treatment | Control Intervention
Number analyzed (Participants) | 25 | 24
Visits to the general practitioner | 1.2 (1.8) | 1.5 (1.7)

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Denominators in the adverse event rates below denote number of participants included in the study analysis excluding ineligible participants.
Arm/Group | Shape-Up Following Cancer Treatment | Control Intervention
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/26 | 3/28
Other Adverse Events (participants affected / at risk) | 0/26 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Shape-Up Following Cancer Treatment (N=26) | Control Intervention (N=28)
Ovarian cancer diagnosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowel obstruction (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes